CLINICAL TRIAL: NCT05342818
Title: Neostigmine Effect on Gastric Residual Volume on Mechanically Ventilated Patients in the Intensive Care Unit. A Comparative Controlled Study by Ondansetron
Brief Title: Evaluating Neostigmine Effect on Reducing Gastric Residual Volume as Compared With Metoclopramide and Ondansetron
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, AHMED ABDELAZIZ SHAMA, LECTURER OF ANESTHESIA AND SURGICAL ICU, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRC112/04/22
Record Dates: First submitted 2022-04-17; First posted 2022-04-25 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Delayed Gastric Emptying
Keywords: gastric residual volume; neostigmine; ondansetron; mechanically ventilated patients
MeSH Terms: conditions — Gastroparesis | interventions — Neostigmine; Ondansetron; Metoclopramide; Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group N (Experimental): patients will receive an intravenous infusion of neostigmine in a dose of 2.5 mg in 100 ml of normal saline within 20 minutes once daily
  Interventions: Drug: Neostigmine; Other: Enteral feeding nutrition; Other: Sequential Organ Failure Assessment (SOFA) score
- Group O (Experimental): patients will receive an intravenous infusion of 8 mg of ondansetron in 100 ml of normal saline once daily for 20 minutes
  Interventions: Drug: Ondansetron 8mg; Other: Enteral feeding nutrition; Other: Sequential Organ Failure Assessment (SOFA) score
- Group M (Experimental): patients will receive metoclopramide in a dose of 10 mg in 100 ml of normal saline once daily for 20 minutes by infusion
  Interventions: Drug: Metoclopramide Injection; Other: Enteral feeding nutrition; Other: Sequential Organ Failure Assessment (SOFA) score

INTERVENTIONS:
Drug: Neostigmine — will be given by infusion in 20 minutes once daily by a nurse blinded to the study drugs
  Other Names: Neostigmine injection
  Arms: Group N
Drug: Ondansetron 8mg — will be given by infusion in 20 minutes once daily by a nurse blinded to the study drugs
  Other Names: Dansetron injection
  Arms: Group O
Drug: Metoclopramide Injection — will be given by infusion in 20 minutes once daily by a nurse blinded to the study drugs
  Other Names: primperan injection
  Arms: Group M
Other: Enteral feeding nutrition — The type and rate of enteral feeding nutrition will be the same for all patients (180ml/3h). All patients have a 30-degree head-up position
  Other Names: Enteral feeding
Other: Sequential Organ Failure Assessment (SOFA) score — SOFA score will be performed on all patients before the beginning of the study
  Other Names: SOFA score

SUMMARY:
One big problem in mechanically ventilated ICU patients is delayed gastric emptying. Delayed gastric emptying in these patients, causes intolerance and high gastric residual volume (GRV) that can lead to abdominal distention, vomiting, increased aspiration risk and consequently increased the length of hospital stay.

In this study, investigators will evaluate Neostigmine's effect in reducing GRV in mechanically ventilated patients and compare its effect with metoclopramide and Ondansetron

.

DETAILED DESCRIPTION:
It has been shown that delayed gastric emptying and high GRV in critically ill patients are associated with increased mortality in these patients. Different kinds of drugs including metoclopramide, erythromycin and cisapride are used, but none of them had conclusive evidence of better eﬀects on each other. Moreover, complications such as dysrhythmia and extrapyramidal side eﬀects limit the use of these drugs.

Another drug that can be used to increase gastric emptying in critically ill patients is neostigmine. Although several studies have evaluated the efficacy of neostigmine on postoperative ileus, very few studies have evaluated the effect of this drug on GRV in ICU patients.

The aim of the current study will be to compare the effects of Neostigmine on gastric residual volume in mechanically ventilated patients in the intensive care unit. A comparative controlled study by Ondansetron.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated ICU patients
* With nasogastric tube feeding
* Gastric Residual Volume >120 mL (3hours after the last gavage)

Exclusion Criteria:

* History of diabetes
* Heart block
* Bradycardia (heart rate <60/min)
* Systolic blood pressure less than 90 mm Hg
* Renal insufficiency
* Using any prokinetic agents such as erythromycin or cisapride within 8 hours before study initiation
* Recent surgery (10 days or less) on the stomach or digestive system
* pregnancy and lactation
* Occurrence of extrapyramidal side effects
* Gastrointestinal (GI) bleeding

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of Gastric Residual Volume(GRV) | 12 hours
  Patients' GRVs will be evaluated before the intervention, then 3, 6, 9 and 12 hours after the intervention using a gavage syringe by an expert nurse who had been unaware of the study groups
Volume of the gastric antrum | 4 days
  After five half-lives of drugs, the volume of the gastric antrum of the patients will be measured by ultrasonography 3 hours after gavage.

SECONDARY OUTCOMES:
Blood albumin | 4 days
  blood sampling daily for four days
Complete Blood Count | 4 days
  blood sampling daily for four days

CONTACTS AND LOCATIONS:
Overall Officials: AHMED A SHAMA, MD, Principal Investigator — Lecturer and consultant of anesthesia and surgical ICU in Tanta University and Faculty of Medicine
Locations (1):
- Sharurah Armed Forces Hospital, Sharurah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No